CLINICAL TRIAL: NCT05843383
Title: Comparison of Ciprofol-based and Propofol-based Total Intravenous Anesthesia on Postoperative Quality of Recovery in Elderly Patients Undergoing Laparoscopic Surgery
Brief Title: Comparison of Ciprofol-based and Propofol-based Total Intravenous Anesthesia on Postoperative Quality of Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY20222308-C-1
Record Dates: First submitted 2023-04-03; First posted 2023-05-06 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-05

CONDITIONS: Anesthetics, Intravenous; Postoperative Complications; Hypnotics and Sedatives; Postoperative Recovery
Keywords: Ciprofol; Propofol
MeSH Terms: conditions — Postoperative Complications | interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; HSK3486; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: participants were anesthetized and were unaware of the grouping. Care providers did not know the grouping. Specific investigators who did the intervention were aware of the grouping. The outcome assessors and the data analyzers did not know the grouping.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciprofol group (Experimental): Ciprofol-based total intravenous anesthesia is given for maintenance of general anesthesia
  Interventions: Drug: Ciprofol
- Propofol group (Experimental): Propofol-based total intravenous anesthesia is given for maintenance of general anesthesia
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Ciprofol — Ciprofol group will be started and maintained total intravenous anesthesia with ciprofol and remifentanil
  Other Names: HSK3486
  Arms: Ciprofol group
Drug: Propofol — Propofol group will be started and maintained total intravenous anesthesia with propofol and remifentanil
  Other Names: 2,6-diisopropylphenol
  Arms: Propofol group

SUMMARY:
Ciprofol is a novel 2,6-disubstituted phenol derivatives and is proved have much higher potency and tighter binding toward ɣ-aminobutyric acid type A (GABAA) receptor while maintaining a fast on-set and recovery time compared to propofol. Except lower incidence of hypotension and respiratory depression, it has no injection pain and infusion syndrome compared with propofol. There is no study to investigate overall postoperative functional recovery in patients receiving total intravenous anesthesia (TIVA) using ciprofol yet. However, according to study, early quality of recovery according to QoR-15 score is associated with one-month postoperative complications after elective surgery. Therefore, the purpose of this study is to determine whether there is any difference in the quality of postoperative recovery between ciprofol-based and propofol-based TIVA in elderly patients undergoing gastrointestinal surgery. The QoR-15 questionnaire score, pain, nausea/vomiting, and the frequency of complications are evaluated and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective laparoscopic surgery under endotracheal intubation and general anesthesia
* American Society of Anesthesiologists (ASA) classification: I to III;
* Age ≥ 60 years, BMI < 30 kg/m2;
* Unconscious speech audiovisual impairment or unable to cooperate;
* Informed consent has been signed.

Exclusion Criteria:

* Taking any sedative, opioid, or sleep aid drugs;
* Psychiatric or neurological disorder;
* Allergic to ciprofol, propofol or soy, or a family history of malignant hyperthermia;
* Severe liver and kidney dysfunction;
* Operation duration < 2 hours;
* Plan to the intensive care unit with tracheal catheter;
* Have participated in this study or other clinical studies.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery(QoR)-15 questionnaire score at postoperative day 1 | Postoperative day 1
  Quality of life will be evaluated using Quality of Recovery(QoR)-15 questionnaire score at postoperative day 1(minimum value: 0, maximum value: 150, the higher the score, the better the result)

SECONDARY OUTCOMES:
Quality of Recovery(QoR)-15 questionnaire score at postoperative day 2 | Postoperative day 2
  Quality of life will be evaluated using Quality of Recovery(QoR)-15 questionnaire score at postoperative day 2 (minimum value: 0, maximum value: 150, the higher the score, the better the result)
Incidence of injection pain | during anesthesia induction
  Record the incidence of injection pain ( yes or no)
Hemodynamic change | During the operation
  Record the mean arterial pressure (MAP) at different points, including before induction, after induction, immediately after intubation, at the beginning of surgery, at the end of anesthesia, immediately after extubation, and before leaving the room
Vasoactive agents | from start of surgery to end of surgery
  Percentage of patients needed vasoactive agents during anesthesia
Tracheal extubation time | From stopping ciprofol or propofol infusion to awake and withdrawal of tracheal tube, approximately 30 minutes
  Time from cessation of main anaesthetics to tracheal extubation
Postoperative sedation score | Immediately after awake，approximately 1 hour after surgery
  Monitored by the sedation scale called Sedation-Agitation Scale (SAS). SAS is a medical scale used to measure the agitation or sedation level of a person.The score ranges from 1 to 7
Postoperative pain score | Immediately after awake, approximately 1 hour after surgery
  postoperative pain score measured by 11-point VAS (Visual Analogue Scale) score (minimum : 0, maximum : 10, the lower the score, the lesser pain)
Postoperative nausea and vomiting | Immediately after awake, approximately 1 hour after surgery
  Postoperative nausea and vomiting will be evaluated by PONV (Post Operative Nausea And Vomiting) score (no : 0, vomit: 4)
First exhaust time | 24 hours after end of surgery, approximately 24 hours
  Record the first exhaust time After the operation
Hospital stay | From end of surgery to discharge from hospital, on an average of 7 days
  days of hospital stay
Postoperative complications | From end of surgery to discharge from hospital, on an average of 7 days
  Various complications occurred during hospitalization
Adverse event | From end of surgery to discharge from hospital, on an average of 7 days
  Percentage of adverse events occurred during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Haopeng Zhang, Study Chair — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qin L, Ren L, Wan S, Liu G, Luo X, Liu Z, Li F, Yu Y, Liu J, Wei Y. Design, Synthesis, and Evaluation of Novel 2,6-Disubstituted Phenol Derivatives as General Anesthetics. J Med Chem. 2017 May 11;60(9):3606-3617. doi: 10.1021/acs.jmedchem.7b00254. Epub 2017 Apr 28. PMID 28430430
- [Background] Bian Y, Zhang H, Ma S, Jiao Y, Yan P, Liu X, Ma S, Xiong Y, Gu Z, Yu Z, Huang C, Miao L. Mass balance, pharmacokinetics and pharmacodynamics of intravenous HSK3486, a novel anaesthetic, administered to healthy subjects. Br J Clin Pharmacol. 2021 Jan;87(1):93-105. doi: 10.1111/bcp.14363. Epub 2020 Aug 3. PMID 32415708
- [Background] Bakhtiari E, Mousavi SH, Gharavi Fard M. Pharmacological control of pain during propofol injection: a systematic review and meta-analysis. Expert Rev Clin Pharmacol. 2021 Jul;14(7):889-899. doi: 10.1080/17512433.2021.1919084. Epub 2021 Jun 1. PMID 33896305
- [Background] Jalota L, Kalira V, George E, Shi YY, Hornuss C, Radke O, Pace NL, Apfel CC; Perioperative Clinical Research Core. Prevention of pain on injection of propofol: systematic review and meta-analysis. BMJ. 2011 Mar 15;342:d1110. doi: 10.1136/bmj.d1110. PMID 21406529
- [Background] Luo Z, Tu H, Zhang X, Wang X, Ouyang W, Wei X, Zou X, Zhu Z, Li Y, Shangguan W, Wu H, Wang Y, Guo Q. Efficacy and Safety of HSK3486 for Anesthesia/Sedation in Patients Undergoing Fiberoptic Bronchoscopy: A Multicenter, Double-Blind, Propofol-Controlled, Randomized, Phase 3 Study. CNS Drugs. 2022 Mar;36(3):301-313. doi: 10.1007/s40263-021-00890-1. Epub 2022 Feb 14. PMID 35157236
- [Background] Campfort M, Cayla C, Lasocki S, Rineau E, Leger M. Early quality of recovery according to QoR-15 score is associated with one-month postoperative complications after elective surgery. J Clin Anesth. 2022 Jun;78:110638. doi: 10.1016/j.jclinane.2021.110638. Epub 2022 Jan 13. PMID 35033845